CLINICAL TRIAL: NCT00112151
Title: Testosterone Supplementation and Exercise in Elderly Men
Brief Title: TEAM: Testosterone Supplementation and Exercise in Elderly Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02-1056; R01AG019339 (NIH)
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: andropause; hypogonadism; AndroGel; exercise; PRT; Testosterone; T supplementation
MeSH Terms: conditions — Hypogonadism; Motor Activity | interventions — Testosterone; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- LowT+Resistance Training (Experimental): Low Dose Testosterone Group applies one 2.5 gm active packet and one placebo packet, titrated to a target blood range of 400-550 pg/ml)
  1 year standard Progressive Resistance Training(PRT) program
  Interventions: Drug: LowT; Behavioral: Resistance Training
- LowT+No Resistance training (Experimental): Low Dose Testosterone Group applies one 2.5 gm active packet and one placebo packet, titrated to a target blood range of 400-550 pg/ml)
  No exercise program
  Interventions: Drug: LowT
- HighT+Resistance Training (Experimental): High Dose Testosterone Group applies two 2.5 gm active packets, titrated to a target blood range of 600-1000 pg/ml)
  1 year standard Progressive Resistance Training(PRT) program
  Interventions: Behavioral: Resistance Training; Drug: HighT
- HighT+No Resistance Training (Experimental): High Dose Testosterone Group applies two 2.5 gm active packets, titrated to a target blood range of 600-1000 pg/ml)
  No exercise program
  Interventions: Drug: HighT
- Placebo+Resistance Training (Active Comparator): Placebo Group applies two 2.5 gm placebo packets
  1 year standard Progressive Resistance Training(PRT) program
  Interventions: Behavioral: Resistance Training; Drug: Placebo
- Placebo+No Resistance Training (Placebo Comparator): Placebo group applies two 2.5 gm placebo packets
  No exercise program
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LowT — Low Dose Testosterone Group applies one 2.5 gm active packet and one placebo packet, titrated to a target blood range of 400-550 pg/ml)during the first 12 weeks. Total exposure duration is 52 weeks.
  Other Names: Androgel
  Arms: LowT+No Resistance training; LowT+Resistance Training
Behavioral: Resistance Training — Weight training 45-60 minutes 3 times per week
  Other Names: PRT; Progressive resistance training
  Arms: HighT+Resistance Training; LowT+Resistance Training; Placebo+Resistance Training
Drug: Placebo — 2.5 gm gel packets applied once daily. Sham adjustments made during the first 12 weeks. Duration is 52 weeks.
  Arms: Placebo+No Resistance Training; Placebo+Resistance Training
Drug: HighT — High Dose Testosterone Group applies two 2.5 gm active packets, titrated to a target blood range of 600-1000 pg/ml)during the first 12 weeks. Total exposure duration is 52 weeks.
  Other Names: Androgel
  Arms: HighT+No Resistance Training; HighT+Resistance Training

SUMMARY:
The purpose of this study is to evaluate the effects of testosterone supplementation (AndroGel) on body composition, strength, endurance, cognition, and function in older men.

DETAILED DESCRIPTION:
Studies suggest that testosterone (T) replacement in healthy elderly men has beneficial effects on body composition, muscle, bone, memory, and behavior, but the risks of chronic treatment, especially on the prostate, heart, and sleep quality, are not entirely clear. Therefore, it is most desirable to supplement into the lowest "effective" range in elderly men. However, the effects of lower than usual replacement T doses have not been well studied. Furthermore, the possible important interaction of exercise to enhance the positive effects of T supplementation, yet mitigate the possible side effects, has not been studied in older men.

This one-year study will enroll 150 men with low-normal to slightly below normal serum total T levels. Participants will be randomized into one of 6 treatment groups to receive T supplementation (AndroGel) of 25mg/day, 50 mg/day or a placebo crossed with progressive resistance training (PRT) exercise 3 times a week versus none. At the end of the study, participants in the exercise-control group will be offered PRT.

Please see link below for updated version of full protocol.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, untrained men 60 years or older with low-normal testosterone levels (200-350ng/dL)
* Must reside in the Denver metro area

Exclusion Criteria:

* Prostate/breast cancer
* Unable to exercise safely
* severe obesity (>34 body mass index [BMI])
* Polycythemia
* Diabetes
* Use of drugs that could affect T levels
* Cognitive dysfunction (MMSE less than 24)
* PSA above the age-adjusted normal level or AUA greater than 19
* Unable to pass stress test due to active CAD

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2005-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Schwartz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] Schwartz RS, Shuman WP, Bradbury VL, Cain KC, Fellingham GW, Beard JC, Kahn SE, Stratton JR, Cerqueira MD, Abrass IB. Body fat distribution in healthy young and older men. J Gerontol. 1990 Nov;45(6):M181-5. doi: 10.1093/geronj/45.6.m181. PMID 2229940
- [Background] Porter MM, Vandervoort AA, Lexell J. Aging of human muscle: structure, function and adaptability. Scand J Med Sci Sports. 1995 Jun;5(3):129-42. doi: 10.1111/j.1600-0838.1995.tb00026.x. PMID 7552755
- [Background] Jolles J, Verhey FR, Riedel WJ, Houx PJ. Cognitive impairment in elderly people. Predisposing factors and implications for experimental drug studies. Drugs Aging. 1995 Dec;7(6):459-79. doi: 10.2165/00002512-199507060-00006. PMID 8601053
- [Background] Davidson JM, Chen JJ, Crapo L, Gray GD, Greenleaf WJ, Catania JA. Hormonal changes and sexual function in aging men. J Clin Endocrinol Metab. 1983 Jul;57(1):71-7. doi: 10.1210/jcem-57-1-71. PMID 6602143
- [Background] Vitiello MV. Sleep disorders and aging: understanding the causes. J Gerontol A Biol Sci Med Sci. 1997 Jul;52(4):M189-91. doi: 10.1093/gerona/52a.4.m189. No abstract available. PMID 9224429
- [Background] Myers BL, Badia P. Changes in circadian rhythms and sleep quality with aging: mechanisms and interventions. Neurosci Biobehav Rev. 1995 Winter;19(4):553-71. doi: 10.1016/0149-7634(95)00018-6. PMID 8684716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from January 2005 through August 2009 of community dwelling men >=60 years of age in the Denver metropolitan area with active attempts to recruit men from all ethnic populations.
Pre-assignment Details: see eligibility criteria
Period: Overall Study
Arm/Group | LowT+Resistance Training | LowT+No Resistance Training | HighT+Resistance Training | HighT+No Resistance Training | Placebo+Resistance Training | Placebo+No Resistance Training
Started | 28 | 28 | 28 | 27 | 28 | 28
Completed | 24 | 23 | 25 | 24 | 22 | 25
Not Completed | 4 | 5 | 3 | 3 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LowT+Resistance Training | LowT+No Resistance Training | HighT+Resistance Training | HighT+No Resistance Training | Placebo+Resistance Training | Placebo+No Resistance Training | Total
Number analyzed (Participants) | 28 | 28 | 28 | 27 | 28 | 28 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 17 | 13 | 16 | 12 | 82
  >=65 years | 16 | 16 | 11 | 14 | 12 | 16 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (7.6) | 65.6 (4.5) | 64.3 (4.6) | 65.3 (5.5) | 64.7 (4.5) | 66.6 (5.4) | 65.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 28 | 28 | 28 | 27 | 28 | 28 | 167
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 28 | 27 | 28 | 28 | 167

OUTCOME MEASURES:

1. Primary Outcome: Physical Function (CS-PFP Total Score)
Description: Continuous-scale physical function performance test (CS-PFP) which comprises 15 everyday tasks requiring upper and lower body strength and flexibility, balance, coordination and endurance. The CS-PFP was developed to measure performance in higher functioning adults with minimal floor or ceiling effects, and is valid, reliable and sensitive to change. Total and domain scores are scaled from 0 to 100, with higher scores indicating better function.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo + No PRT: Placebo gel; no exercise
- Placebo + PRT: Placebo gel plus progressive resistance training
- Any T + No PRT: T gel supplementation (lower or higher-range); no exercise
- Any T + PRT: T gel supplementation (lower or higher-range) plus progressive resistance training
Arm/Group | Placebo + No PRT | Placebo + PRT | Any T + No PRT | Any T + PRT
Number analyzed (Participants) | 25 | 22 | 47 | 49
units on a scale | 3.1 (6.7) | 3.6 (8.0) | 0.8 (7.3) | 3.3 (7.4)
Statistical Analysis 1: Comparison: Placebo + PRT vs Any T + PRT; As prespecified, the lower- and higher-range T groups were combined (any T). The primary analysis was conducted in the PRT groups and compared CS-PFP at 12 months with any T to placebo, adjusted for baseline CS-PFP score; Test type: Superiority or Other; p < 0.025, Regression, Linear — A one-sided P-value of <0.025 was used to define statistical significance
Statistical Analysis 2: Comparison: Placebo + No PRT vs Any T + No PRT; As prespecified, the lower- and higher-range T groups were combined (any T). To address whether the effects of any T on physical function are the same without PRT, the analysis was also conducted in the No PRT groups, comparing CS-PFP at 12 months with any T to placebo, adjusted for baseline CS-PFP score; Test type: Superiority or Other; p < 0.025, Regression, Linear — A one-sided P-value of <0.025 was used to define statistical significance

2. Secondary Outcome: Upper Body Muscle Strength (1-RM, kg)
Description: The maximal weight a participant could lift once (1-repetition maximum, 1-RM) was assessed at baseline and 12 months. The average of the difference from baseline in 4 upper-body 1-RM measures (bench press,incline press, overhead pull-down, and seated row) are represented.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Any T + No PRT: T gel supplementation (lower- or higher-range); no exercise
- Any T + PRT: T gel supplementation (lower- or higher-range) plus progressive resistance training
Arm/Group | Placebo + No PRT | Placebo + PRT | Any T + No PRT | Any T + PRT
Number analyzed (Participants) | 25 | 22 | 47 | 49
kg | 4.3 (7.7) | 25.5 (11.3) | 7.8 (6.9) | 24.3 (11.6)
Statistical Analysis 1: Comparison: Placebo + PRT vs Any T + PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in average upper body strength with any T to placebo in subjects assigned to PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Placebo + No PRT vs Any T + No PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in average upper body strength with any T to placebo in subjects assigned to no PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear

3. Secondary Outcome: Lower Body Muscle Strength (1-RM, kg)
Description: The maximal weight a participant could lift once [1-repetition maximum, 1-RM] was assessed at baseline and 12 months. The average of the difference from baseline in 3 lower-body 1-RM measures (knee extension, knee flexion, and seated leg press)) are represented.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo + No PRT | Placebo + PRT | Any T + No PRT | Any T + PRT
Number analyzed (Participants) | 25 | 22 | 47 | 49
kg | 9.4 (11.6) | 27.0 (17.0) | 10.5 (10.9) | 28.0 (19.7)
Statistical Analysis 1: Comparison: Placebo + PRT vs Any T + PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in average lower body strength with any T to placebo in subjects assigned to PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Placebo + No PRT vs Any T + No PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in average lower body strength with any T to placebo in subjects assigned to no PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear

4. Secondary Outcome: Power (Power Rig, Watts)
Description: Leg extensor power was evaluated using a Nottingham leg extensor power rig (watts).
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Placebo + No PRT | Placebo + PRT | Any T + No PRT | Any T + PRT
Number analyzed (Participants) | 25 | 22 | 47 | 49
Watts | 4.5 (34.6) | 24.3 (62.0) | 0.8 (36.9) | 5.1 (51.1)
Statistical Analysis 1: Comparison: Placebo + PRT vs Any T + PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in leg extensor power with any T to placebo in subjects assigned to PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Placebo + No PRT vs Any T + No PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in leg extensor power with any T to placebo in subjects assigned to no PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear

5. Secondary Outcome: Fat Mass (kg)
Description: Total change in Fat mass (kg) as evaluated by DXA
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo + No PRT | Placebo + PRT | Any T + No PRT | Any T + PRT
Number analyzed (Participants) | 25 | 22 | 47 | 49
kg | 0.7 (2.3) | -0.6 (1.7) | -1.0 (2.3) | -1.8 (2.5)
Statistical Analysis 1: Comparison: Placebo + PRT vs Any T + PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in fat mass measured by dual x-ray absorptiometry (DXA) with any T to placebo in subjects assigned to PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Placebo + No PRT vs Any T + No PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in fat mass measured by dual x-ray absorptiometry (DXA) with any T to placebo in subjects assigned to no PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear

6. Secondary Outcome: Fat Free Mass (kg)
Description: Total change in Fat free mass (kg) as evaluated by DXA
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo + No PRT | Placebo + PRT | Any T + No PRT | Any T + PRT
Number analyzed (Participants) | 25 | 22 | 47 | 49
kg | 0.1 (1.7) | 0.4 (2.1) | 1.0 (2.2) | 2.1 (2.4)
Statistical Analysis 1: Comparison: Placebo + PRT vs Any T + PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in fat free mass measured by dual x-ray absorptiometry (DXA) with any T to placebo in subjects assigned to PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Placebo + No PRT vs Any T + No PRT; As prespecified, the lower- and higher-range T groups were combined (Any T). The analysis compared change from baseline to 12 months in fat free mass measured by dual x-ray absorptiometry (DXA) with any T to placebo in subjects assigned to no PRT; Test type: Superiority or Other; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 1 year
Description: Systematic assessments were done at baseline, 4, 12, 26 and 52 weeks. As prespecified, adverse events were analyzed according to T dosing (e.g. placebo, lower-range T, and higher-range T).
Groups:
- Placebo: Placebo gel with or without progressive resistance training
- Lower-range T: T gel supplementation targeting a total serum T concentration of 400-550ng/dL, with our without progressive resistance training
- Higher-range T: T gel supplementation targeting a total serum T concentration of 600-1000ng/dL, with our without progressive resistance training
Arm/Group | Placebo | Lower-range T | Higher-range T
Serious Adverse Events (participants affected / at risk) | 30/47 | 33/47 | 38/49
Other Adverse Events (participants affected / at risk) | 23/47 | 14/47 | 25/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Lower-range T (N=47) | Higher-range T (N=49)
Total serious cardiovascular adverse events (Cardiac disorders) | 10 (11) | 2 (3) | 1 (1) — Includes acute coronary syndrome, arrhythmia, aortic aneurysm, syncope/presyncope
Other noncardiovascular serious adverse events (General disorders) | 20 (53) | 31 (55) | 37 (64)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | Lower-range T (N=47) | Higher-range T (N=49)
Persistently elevated HCT >= 54% (Blood and lymphatic system disorders) | 3 (3) | 2 (4) | 11 (13) — Polycythemia or persistent elevated hematocrit >= 54%
Persistently elevated PSA (Renal and urinary disorders) | 9 (14) | 5 (9) | 7 (13) — Persistent elevated PSA representing an increase of >=0.75 ng/mL over baseline
Elevated AUA (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) — American Urological Association (AUA) BPH Symptom Score Index >= 20
Persistently elevated liver function tests (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) — Alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of normal
Daytime somnolence/hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) — Somnolence = Epworth Sleepiness Score > 16; hypoxia is daytime arterial oxygen saturation by pulse oximetry < 88%
Other nonserious adverse events (General disorders) | 9 (12) | 6 (6) | 7 (7) — Other nonserious adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No